CLINICAL TRIAL: NCT06240104
Title: A Randomized Controlled Study on Continuous Monitoring of Cardiac Index Variability to Guide Patients With Perioperative Myocardial Injury to Wean From Mechanical Ventilation
Brief Title: Monitoring of Heart to Guide Myocardial Injury Patients to Wean From Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Shu, associate professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDL2023-09
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Myocardial Ischaemia During Surgery
Keywords: cardiac index variability; wean from mechanical ventilation; perioperative myocardial injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CI group (Experimental): the cardiac index (CI) is continuously monitored during the weaning process
  Interventions: Diagnostic Test: cardiac output index monitor
- control group (No Intervention): No intervention measures

INTERVENTIONS:
Diagnostic Test: cardiac output index monitor — During the spontaneous breathing test phase, the cardiac index (CI) is continuously monitored from 15-30 minutes prior to the start of the test. Patients who have successfully completed the spontaneous breathing test and increased their CI by more than 30% and meet ordinary weaning indications can have their tracheal intubation removed.
  Arms: CI group

SUMMARY:
The goal of this prospective randomized controlled clinical trail is to explore the value of integrating continuous cardiac index variability indicators with existing weaning standards to guide perioperative myocardial injury patients weaning. The main question it aims to answer is: whether the introduction of new indicators for weaning standards can improve the success rate of weaning. Treatment that'll be given to participants is: the cardiac index (CI) is continuously monitored from 15-30 minutes prior to the start of the weaning from ventilation. Participants who increase their CI by more than 30% can have their tracheal intubation removed. Researchers will compare the weaning success rate of CI group and control group.

DETAILED DESCRIPTION:
In this study, investigator'll recruit participants of perioperative myocardial injury as the research objects, the continuous cardiac index variability index was added to the current traditional weaning standard to form a new weaning standard. In this prospective, randomized, and controlled study, the impact of the new weaning standard and the traditional weaning standard on weaning failure rate was compared. Whether the new weaning standard is superior to ordinary weaning standards is evaluated in terms of participants prognosis, incidence of complications, and medical resource consumption.

Quality assurance plan that addresses data validation and registry procedures: Two researchers who have received unified training record and register participant data separately, and a third researcher conducts weekly data checks to compare data entered into the registry against predefined rules for range. The source data will be verified to assess the accuracy, completeness of registry data by comparing the data to medical records and paper or electronic case report forms.

Standard Operating Procedures to address participant recruitment, data collection, data management, data analysis, reporting for adverse events, and change management will be formulated before recruit.

The estimation of sample size is based on testing that the new weaning standard is superior to traditional standards in improving weaning success rate. According to previous reports and our previous study data, the sample size was calculated using PASS 11.0 software. The results showed that 91 cases were needed in each group. Considering a 5% dropout rate, 100 participants were included in each group for a total of 200 participants.

Plan for missing data: Investigator will verify the data monthly and recruit sufficient participants according to the research protocol and statistical requirements.

Statistical analysis plan:

* Use SAS 10.0 statistical software for statistical analysis. Quantitative data is represented by mean, standard deviation, median and interquartile range, while count data is represented by absolute frequency and composition ratio.
* The comparison of weaning success rates for primary study endpoints was conducted using the confidence interval method. Calculate the one-sided 95% confidence interval for the difference in success rates between the new offline standard group and the traditional offline standard group, if this interval is greater than δ Value, it can be considered that the new offline standard is superior to the traditional offline standard.
* Secondary study endpoints: basic demographic characteristics and clinical indicators, postoperative mechanical ventilation time, ICU stay, hospital stay, and incidence of ventilator-associated pneumonia. Student t-tests and rank sum tests were used for inter group comparison of quantitative data; The inter group comparison of counting data adopts kapa Inspection. All tests are bilateral tests with significance levels α = 0.05.
* The patient's survival status was described using Kaplan Meier survival curves, and intergroup differences were tested using the Breslow method.

ELIGIBILITY:
Inclusion Criteria:

* Perioperative myocardial injury patients
* Age>18 years;
* Acute Physiology and Chronic Health Evaluation II (APACHEII)>8 ;
* The weaning process has not yet started after surgery;
* Expected postoperative cumulative mechanical ventilation time>24 hours.

Exclusion Criteria:

* Pregnancy or childbirth less than 42 days;
* Patients and their families are unable to cooperate with treatment;
* The cumulative actual mechanical ventilation time after surgery is ≤ 24 hours;
* Interruption of mechanical ventilation treatment due to death or other reasons before entering the weaning process;
* Patients who retain artificial airways after weaning;
* Patients who plan to start non-invasive mechanical ventilation treatment immediately after weaning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
weaning success rate | through study completion, an average of 1 year

SECONDARY OUTCOMES:
in-ICU mortality | through study completion, an average of 1 year
28 day mortality | through study completion, an average of 1 year
The incidence of ventilator-associated pneumonia | through study completion, an average of 1 year
length of stay in ICU | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 year after publication, for 1 years
Access Criteria: The project leader can be contacted to obtain the original data under reasonable and legal conditions.